CLINICAL TRIAL: NCT05678855
Title: The Effect of multımedıa-based educatıon ın dıstance learnıng on nursıng Students' academıc Success and motıvatıon: A randomızed Controlled Study
Brief Title: The Effect of multımedıa-based educatıon ın dıstance learnıng on nursıng Students'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Esin Cetinkaya Uslusoy, Associate Professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EsinMultimedia
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Nursing Students
Keywords: multimedia based education

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: students were given information about the study, but not in which group they are included. Thus, blinding was ensured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Control Group: The topics of the course were prepared by the researcher using PowerPoint. Before starting the courses, it is ensured that all students attended the course using the Microsoft Teams program. The contents prepared were presented to the students in the control group with the traditional education method on a weekly basis.
- experimental group (Experimental): a) Experimental Group: First, the topics of the course were prepared by the researcher using multimedia tools. Before starting the courses, it is ensured that all students attended the course using the Microsoft Teams program. The contents prepared were presented to the students in the experimental group in an interactive way on a weekly basis.
  Interventions: Behavioral: A randomızed Controlled Study with pre-test and post-test

INTERVENTIONS:
Behavioral: A randomızed Controlled Study with pre-test and post-test — The intervention in this study is to apply multimedia-based instruction in distance education to the experimental group. control group students received distance education through traditional teaching. Experimental group students received distance education through interactive teaching prepared with multimedia tools. Experimental group, interactions were made using applications such as Icebreaker, Puzzle, QR code, Mentimeter, and Padlet. In addition, animation, infographics, animated slides (Multimedia tools) were used for the experimental group.In the control group, plain narration was given. Tests were administered to both groups before and after the intervention.
  Arms: experimental group

SUMMARY:
Abstract Objective: In this study, it is aimed to evaluate the effect of multimedia teaching materials on students' academic achievement and motivation in teaching nursing process course.

Design: Randomized controlled trial. Settings: Public university. Participants: The research was carried out on first year nursing students (N=70).

Methods: Data; were collected using the introductory features form, academic achievement evaluation (quiz) and Instructional Materials Motivation Questionnaire. Research data were collected using online questionnaires. The experimental group students were presented with the contents of the nursing process course, which was prepared with multimedia materials for two hours in seven weeks with distance education. The control group students were taught by distance education and traditional lectures for two hours in seven weeks.

DETAILED DESCRIPTION:
This research was carried out in an experimental design with a pre-test-post-test control group to examine the effect of using multimedia instructional materials in the teaching of the Nursing Process course, which is a theoretical course given by the distance learning method, on academic success and motivation of the students. The course presentations in the research were presented to the students with the Microsoft Teams program. Data collection was carried out by the researcher via Google Forms.

Participants and Setting The participants of this study are first-year students studying at the Department of Nursing at a state university (N=70).

Procedures Within the scope of this study, the Nursing Process course was created as an elective course. The elective course of the Nursing Process is taught for 14 weeks as two hours per week using theoretical and case presentation methods. The first seven-week topics consist of general information about the Nursing Process (such as its history, importance, and steps). In the next seven weeks, students present examples of the Nursing Process to the class. This research was carried out in the first seven weeks when the theoretical subjects were given. Students who chose this course are listed. The students who volunteered to participate in the study were divided into two groups: the experimental group and the control group (see randomization). This course was given to both groups for 2 hours per week for seven weeks. The course duration is limited to approximately 40-45 minutes.

The Nursing Process course was prepared with multimedia tools through the Microsoft Teams program in distance learning and presented to the experimental group with content appealing to many senses. The control group, on the other hand, was given by traditional narration through the Microsoft Teams program in distance learning. In data collection, a sociodemographic characteristics survey and instructional materials motivation survey were applied to the students in both groups before the intervention. After the attempt, all of the students were evaluated for academic success (Quiz). Instructional materials motivation survey was applied to the groups for the second time.

Interventions

Groups received the same theoretical content for seven weeks. However, there are differences between the groups in terms of the presentation of the course. The content acquisition activities of the groups are divided as follows:

1. Experimental Group: First, the topics of the course were prepared by the researcher using multimedia tools. Before starting the courses, it is ensured that all students attended the course using the Microsoft Teams program. The contents prepared were presented to the students in the experimental group in an interactive way on a weekly basis.
2. Control Group: The topics of the course were prepared by the researcher using PowerPoint. Before starting the courses, it is ensured that all students attended the course using the Microsoft Teams program. The contents prepared were presented to the students in the control group in an interactive way with the traditional education method on a weekly basis.

In addition to theoretical activities for content acquisition, interactions are available for both groups. Interactions in the control group were provided by the question and answer method. In the experimental group, interactions were made using applications such as Icebreaker, Puzzle, QR code, Mentimeter, and Padlet.

Preparation of Multimedia Instructional Materials Used in the Nursing Process Course created for the experimental group Instruments

Sociodemographic characteristics form, academic success assessment (quiz), and Instructional Materials Motivation Survey were used to collect the data of the study. Surveys are given below:

* Sociodemographic Characteristics Form - data were collected including age, gender, the status of choosing the nursing department, whether they previously received distance learning, and their status of gaining professional knowledge through distance learning.
* Academic Success Assessment (Quiz) - It is a 20-question quiz created by the researcher to measure the success of the students in the Nursing Process course. The duration of this exam is 20 minutes and each question is worth 5 points. This was conducted as an online exam in the University's teaching management system.
* Instructional Materials Motivation Survey (IMMS) - Instructional Materials Motivation Survey was prepared by J. M. Keller (2009) as a motivation model for attention, relevance, confidence, and satisfaction (Attention, Relevance, Confidence, Satisfaction-ARCS Model). The Turkish validity and reliability study of the Instructional Materials Motivation Survey (IMMS) was conducted by Hulya Kutu and Mustafa Sozbilir (2011). IMMS identifies changes in students' motivation when faced with instructional materials based on key components (attention, relevance, confidence, and satisfaction). As a result of the analyzes, the survey was adapted to Turkish with two factors and 24 items. The reliability (Cronbach's Alpha) internal consistency coefficient of the survey was found to be 0.83 for the total survey, and 0.79 and 0.69 for the sub-factors, respectively. The sub-dimensions of the scale are divided into attention-relevance and confidence-satisfaction. Items of the scale are attention-relevance (11) "When I first learned about the content, I saw that there were some interesting things in this course that caught my attention."; confidence-satisfaction (13) "I enjoyed the course". The scale is in the type of self-report. The survey is a 5-point Likert type (1 = Totally disagree, 5 = Totally agree). The lowest score that can be obtained from the scale is 24, and the highest score is 120. The higher the total score, the stronger the motivation to learn. In this study, Cronbach's alpha value of the Instructional Materials Motivation Survey was found to be 0.92; it was 0.86 for the attention-relevance sub-dimension, and 0.82 for the confidence-satisfaction sub-dimension.

Randomization The sample consisted of first-year students (N=70) who chose the "Nursing Process" elective course in the spring semester. All students agreed to participate in the study. Students were listed for randomization, each student was given a number, and a random assignment was made to the experimental (N=38) and control groups (N=32) with the help of a computer program (www.random.org).

Ethics committee approval was received for the study from Suleyman Demirel Universty.

ELIGIBILITY:
Inclusion Criteria:

* Students who had internet access and volunteered to participate were included in the study.

Exclusion Criteria:

* Students who did not have internet access and did not volunteer to participate were not included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Characteristics Form | one week
  data were collected including age, gender, the status of choosing the nursing department, whether they previously received distance learning, and their status of gaining professional knowledge through distance learning.
Academic Success Assessment (Quiz) | 8th week
  It is a 20-question quiz created by the researcher to measure the success of the students in the Nursing Process course. The duration of this exam is 20 minutes and each question is worth 5 points. This was conducted as an online exam in the University's teaching management system.
Instructional Materials Motivation Survey (IMMS) | 8 weeks
  Instructional Materials Motivation Survey was prepared by J. M. Keller (2009) as a motivation model for attention, relevance, confidence, and satisfaction. IMMS identifies changes in students' motivation when faced with instructional materials based on key components. As a result of the analyzes, the survey was adapted to Turkish with two factors and 24 items. The reliability (Cronbach's Alpha) internal consistency coefficient of the survey was found to be 0.83 for the total survey, and 0.79 and 0.69 for the sub-factors, respectively. The sub-dimensions of the scale are divided into attention-relevance and confidence-satisfaction. The scale is in the type of self-report. The survey is a 5-point Likert type (1 = Totally disagree, 5 = Totally agree). The lowest score that can be obtained from the scale is 24, and the highest score is 120. The higher the total score, the stronger the motivation to learn.

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCoy L, Lewis JH, Dalton D. Gamification and Multimedia for Medical Education: A Landscape Review. J Am Osteopath Assoc. 2016 Jan;116(1):22-34. doi: 10.7556/jaoa.2016.003. PMID 26745561